CLINICAL TRIAL: NCT05370248
Title: The Effect of 6 ml/kg vs 10 ml/kg Tidal Volume on Diaphragm Dysfunction in Critically Mechanically Ventilated Patient: a Randomized Clinical Trial
Brief Title: The Effect of 6 ml/kg vs 10 ml/kg Tidal Volume on Diaphragm Dysfunction in Critically Mechanically Ventilated Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Darma Putra Sitepu, Anesthesiologist Consultant In-Training, Principal Investigator, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DPS1
Record Dates: First submitted 2022-04-28; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Mechanical Ventilation Complication
Keywords: Mechanical ventilation; Diaphragm dysfunction
MeSH Terms: interventions — Tidal Volume

STUDY DESIGN:
Intervention Model Description: Patient was divided into group A and B. Group A received tidal volume of 6 ml/kg and group B received tidal volume of 10 ml/kg.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blinded to which group they belong and they have given consent to that.
  The person assigning patients to each group is the research assistant. The person setting the mechanical ventilator is the anesthesiology resident. The person assessing outcome with ultrasound is radiology department staff, who does not know which group the patient belong.
  The person assessing outcome of interleukin is laboratory personnel, who does not know which group the patient belong.
  The person collecting and freezing data into worksheet is the research assistant.
  The person analyzing final data is the primary investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The six (Experimental): The group who received tidal volume of 6 ml/kg from mechanical ventilation
  Interventions: Other: Tidal volume 6 ml/kg
- The ten (Active Comparator): The group who received tidal volume of 10 ml/kg from mechanical ventilation
  Interventions: Other: Tidal volume 10 ml/kg

INTERVENTIONS:
Other: Tidal volume 6 ml/kg — Tidal volume is defined as the amount of air that moves in or out of the lungs with each respiratory cycle, given by the mechanical ventilator.
  Arms: The six
Other: Tidal volume 10 ml/kg — Tidal volume is defined as the amount of air that moves in or out of the lungs with each respiratory cycle, given by the mechanical ventilator.
  Arms: The ten

SUMMARY:
This is a randomized clinical trial to measure the effect of tidal volume (group 6 ml/kg vs 10 ml/kg) on diaphragm dysfunction on mechanically ventilated critical patient.

DETAILED DESCRIPTION:
Patient was enrolled in the first day receiving mechanical ventilation in ICU. Patient was included to group A or group B. Group A patient will receive tidal volume of 6 ml/kg and group B patient will receive tidal volume of 10 ml/kg. The assignment was randomized. Followed for 3 days. After 24, 48, and 72 hours, patient blood will be collected to measure the interleukin value, and diaphragm dysfunction will be observed by the use of ultrasonography by expert doctor from radiology department. Data will be analyzed statistically if there is an effect of tidal volume difference on diaphragm dysfunction and interleukin-6 as marker of inflammation. The minimal sample of patient is 44 patients.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years old
* Critically ill patients

Exclusion Criteria:

* Patient with ARDS (PaO2/FiO2 <200)
* Pregnant woman
* Patient with history of cardiac or thorax surgery 14 days prior to admission
* Patient with severe peripheral musculoskeletal conditions
* Patient with prolonged in-hospital stay (>2 weeks) in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
DD-24 | 24 hours after mechanical ventilation
  Diaphragm dysfunction 24 hours after mechanical ventilation assessed by ultrasound.
DD-48 | 48 hours after mechanical ventilation
  Diaphragm dysfunction 48 hours after mechanical ventilation assessed by ultrasound.
DD-72 | 72 hours after mechanical ventilation
  Diaphragm dysfunction 72 hours after mechanical ventilation assessed by ultrasound.

SECONDARY OUTCOMES:
IL-6-24 | 24 hours after mechanical ventilation
  Blook interleukin 6 24 hours after mechanical ventilation
IL-6-48 | 48 hours after mechanical ventilation
  Blook interleukin 6 48 hours after mechanical ventilation
IL-6-72 | 72 hours after mechanical ventilation
  Blook interleukin 6 72 hours after mechanical ventilation

OTHER OUTCOMES:
Discharge outcome | Up to three months after mechanical ventilation
  The outcome at hospital discharge (alive or death)
LOS in hospital | Up to three months after mechanical ventilation
  Length of stay (days) in hospital
LOS in ICU | Up to three months after mechanical ventilation
  Length of stay (days) in ICU
Weaning failure | Up to three months after mechanical ventilation
  The condition where patient failed for spontaneous breathing trial after mechanical ventilation. Grouped into success/failed.
Intubation time | At extubation after mechanical ventilation
  Time (hours) long when a patient was intubated

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, Dr, Study Chair — Dr Cipto Mangunkusumo Hospital
Locations (1):
- Dr Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared since it is belong to the hospital and patient did not consent it to be published.

REFERENCES:
- [Background] Mehta AB, Syeda SN, Wiener RS, Walkey AJ. Epidemiological trends in invasive mechanical ventilation in the United States: A population-based study. J Crit Care. 2015 Dec;30(6):1217-21. doi: 10.1016/j.jcrc.2015.07.007. Epub 2015 Jul 16. PMID 26271686
- [Background] Tremblay LN, Slutsky AS. Ventilator-induced lung injury: from the bench to the bedside. Intensive Care Med. 2006 Jan;32(1):24-33. doi: 10.1007/s00134-005-2817-8. Epub 2005 Oct 18. No abstract available. PMID 16231069
- [Background] Brochard L, Slutsky A, Pesenti A. Mechanical Ventilation to Minimize Progression of Lung Injury in Acute Respiratory Failure. Am J Respir Crit Care Med. 2017 Feb 15;195(4):438-442. doi: 10.1164/rccm.201605-1081CP. PMID 27626833
- [Background] Petrof BJ. Diaphragm Weakness in the Critically Ill: Basic Mechanisms Reveal Therapeutic Opportunities. Chest. 2018 Dec;154(6):1395-1403. doi: 10.1016/j.chest.2018.08.1028. Epub 2018 Aug 23. PMID 30144420
- [Background] Supinski GS, Morris PE, Dhar S, Callahan LA. Diaphragm Dysfunction in Critical Illness. Chest. 2018 Apr;153(4):1040-1051. doi: 10.1016/j.chest.2017.08.1157. Epub 2017 Sep 5. PMID 28887062
- [Background] Demoule A, Jung B, Prodanovic H, Molinari N, Chanques G, Coirault C, Matecki S, Duguet A, Similowski T, Jaber S. Diaphragm dysfunction on admission to the intensive care unit. Prevalence, risk factors, and prognostic impact-a prospective study. Am J Respir Crit Care Med. 2013 Jul 15;188(2):213-9. doi: 10.1164/rccm.201209-1668OC. PMID 23641946
- [Background] Zambon M, Greco M, Bocchino S, Cabrini L, Beccaria PF, Zangrillo A. Assessment of diaphragmatic dysfunction in the critically ill patient with ultrasound: a systematic review. Intensive Care Med. 2017 Jan;43(1):29-38. doi: 10.1007/s00134-016-4524-z. Epub 2016 Sep 12. PMID 27620292
- [Background] Moxham J, Goldstone J. Assessment of respiratory muscle strength in the intensive care unit. Eur Respir J. 1994 Nov;7(11):2057-61. PMID 7875282